CLINICAL TRIAL: NCT06218394
Title: Comparison of Microneedling vs. Autologous Concentrated Growth Factor for the Treatment of Female Androgenetic Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230984
Record Dates: First submitted 2024-01-02; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-12

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Percutaneous Collagen Induction; Minoxidil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- microneedling (Experimental)
  Interventions: Procedure: microneedling
- autologous concentrated growth factor (Experimental)
  Interventions: Procedure: Autologous Concentrated Growth Factor
- 5% minoxidil (Active Comparator)
  Interventions: Drug: 5% minoxidil

INTERVENTIONS:
Procedure: microneedling — The microneedling technique (Electric microneedle, F6, China Bohui Meicui Bioengineering Technology Guangzhou Co., LTD.) performed in the targeted areas using a sterile micro needles stamp. In this study, the needle length was adjusted to 0.7~1 mm according to the grade of hair loss and the degree of tolerance of the patient. Before microneedling treatment, the scalp was disinfected with 75% alcohol, and then 1 ml of nutritional dressing for the scalp was applied externally, and the microneedle pen was gently touched to the scalp vertically for pricking. Patients are instructed to refrain from shampooing, warm baths, and strenuous exercise for 8 hours after treatment. Each patient was treated by microneedling once every 2 weeks for a total of 12 treatments.
  Arms: microneedling
Procedure: Autologous Concentrated Growth Factor — 1. 27~36ml of autologous venous blood is collected in a sterile Vacuette tube without anticoagulant solution, and centrifuged by Medifuge variable speed centrifuge (Silfradent company, Italy) for about 13min (accelerated for 30s; 2700 r/min, 2 min; 2400 r/min, 4min; 2700r/min, 4min; 3300r/min, 3 min; decelerated for 36s to stop). The lowest layer retains 2.5ml of CGF per 9ml of venous blood.
  2. The scalp is cleaned, disinfected and anesthetized, CGF is extracted with a 2.5ml syringe, and the disposable sterile needle roller handle is slowly rolled in the hair loss area, and the CGF is applied to the corresponding scalp part for introduction treatment while rolling, and the force is uniform and stable, repeating back and forth several times, to the extent that the patient can tolerate and the skin in the treatment area is slightly red. The operation time is about 15~20 minutes.
  Arms: autologous concentrated growth factor
Drug: 5% minoxidil — topical 5% minoxidil, 1 ml, once daily
  Arms: 5% minoxidil

SUMMARY:
Microneedling and autologous concentrated growth factor (CGF) have established their potential effect in inducing hair regrowth. No study has compared the effect of microneedling and CGF in the treatment of female androgenetic alopecia (AGA).

DETAILED DESCRIPTION:
Microneedling is a minimally invasive technique consisting of sterile microneedles for repetitive cutaneous puncturing that increase hair regrowth by growth factor release. Concentrated growth factor (CGF) is a form of platelet concentrate (PC) and concentrates higher levels of growth factors because of its varying programmed centrifugation process. Previous studies have showed that CGF injection in hairless scalp could enhance the hair density and optimize the hairless appearance in AGA patients. Both microneedling and CGF have established their potential effect in inducing hair regrowth. No study has compared the effect of microneedling and CGF in the treatment of female androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 years;；
2. clinical diagnosis of female pattern hair loss；
3. no previous laser treatments for AGA in the past six months before enrollment； 4) willingness to provide pictures and follow-up studies.

Exclusion Criteria:

1. if presented with severe diseases of internal organs, eyes, or skin;
2. inflammation, infection, or unhealed wounds on the skin around the site of treatment on the head;
3. systematic treatment with corticosteroids or other immunosuppressants and immunomodulators in the past 3 months.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
TAHC | week 24
  Use the trichoscopy to assess the changing number of non-vellus hairs in the target area .

SECONDARY OUTCOMES:
HGQA | week 8, week 12, week 16, week 24, week 36
  Hair growth questionnaire assessment
TAHC | week 8, week 12, week 20, week 36
  Use the trichoscopy to assess the changing number of non-vellus hairs in the target area
TAHW | week 8, week 12, week 16, week 24, week 36
  Use the trichoscopy to assess the changing diameter of non-vellus hairs in the target area
IGA | week 8, week 12, week 16, week 24, week 36
  Investigator's Global Assessment. IGA was evaluated using a 7-point scale as follows: -3= obvious reduction of hair; -2= moderate reduction of hair; -1= mild reduction of hair; 0= change; 1= mild growth of hair; 2= moderate growth of hair; 3= obvious growth of hair.
Grade of Ludwig and Norwood-Hamilton Classification | week 12, week 24, week 36
  The Grade of Ludwig and Norwood-Hamilton Classification
SSA | week 8, week 12, week 16, week 24, week 36
  Subject self-assessment. SSA was evaluated using a 7-point scale as follows: -3= obvious reduction of hair; -2= moderate reduction of hair; -1= mild reduction of hair; 0= change; 1= mild growth of hair; 2= moderate growth of hair; 3= obvious growth of hair.

OTHER OUTCOMES:
Incidents of adverse events | through study completion, an average of 36 weeks
  Safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Xianjie Wu, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are not publicly available due to the privacy of research participants but are available from the sponsor upon reasonable request.